CLINICAL TRIAL: NCT05186753
Title: A Multi-Part, Randomized, Double-Blind, Placebo-Controlled Phase 2 Clinical Study of The Safety and Efficacy of CGT9486 in Subjects With Nonadvanced Systemic Mastocytosis
Brief Title: (Summit) A Study to Evaluate the Efficacy and Safety of CGT9486 Versus Placebo in Patients With Indolent or Smoldering Systemic Mastocytosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CGT9486-21-202
Record Dates: First submitted 2021-11-19; First posted 2022-01-11 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: SSM; Mastocytosis, Indolent; Mastocytosis, Systemic; Mastocytosis; ISM; BMM; Smoldering Systemic Mastocytosis; Bone Marrow Mastocytosis
Keywords: Systemic Mastocytosis; Immune Complex Diseases; Immune System Diseases; Hypersensitivity; Hematologic Diseases; NonAdvSM; D816V; KIT D816V; Bezuclastinib; CGT9486; CGT; PLX; Nonadvanced Systemic Mastocytosis; PLX9486; Indolent Systemic Mastocytosis; ISM; Smoldering Systemic Mastocytosis; BMM; Bone Marrow Mastocytosis; SSM
MeSH Terms: conditions — Mastocytosis; Mastocytosis, Systemic; Immune Complex Diseases; Immune System Diseases; Hypersensitivity; Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: In Part 1a and 1b of the study, patients with NonAdvSM will be randomly assigned to 1 of 2 dose levels of bezuclastinib plus BSC, or to placebo plus BSC. Upon analysis of the Part 1 data, a dose will be selected for Part 2. In Part 2, patients with NonAdvSM will be randomly assigned to the selected dose of bezuclastinib plus BSC, or to placebo plus BSC.
  Patients who complete Part 1 or Part 2 may participate in Part 3 in which all patients will receive bezuclastinib plus BSC.
  Subjects participating in the substudy will receive open-label bezuclastinib plus BSC.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- (Part 1a) Bezuclastinib Dose 1 + BSC (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation A)
- (Part 1a) Bezuclastinib Dose 2 + BSC (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation A)
- (Part 1a) Placebo + BSC (Placebo Comparator)
  Interventions: Drug: Placebo Tablets
- (Part 1b) Bezuclastinib Dose 1 + BSC (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation B)
- (Part 1b) Bezuclastinib Dose 2 + BSC (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation B)
- (Part 1b) Placebo + BSC (Placebo Comparator)
  Interventions: Drug: Placebo Tablets
- (Part 2) Bezuclastinib Selected Dose + BSC (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation B)
- (Part 2) Placebo + BSC (Placebo Comparator)
  Interventions: Drug: Placebo Tablets
- (Part 3) Bezuclastinib + BSC (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation A); Drug: Bezuclastinib Tablets (Formulation B)
- (Prior Therapy Sub-study) Bezuclastinib (Experimental)
  Interventions: Drug: Bezuclastinib Tablets (Formulation B)

INTERVENTIONS:
Drug: Bezuclastinib Tablets (Formulation A) — Bezuclastinib will be administered orally, once daily continuously for 28-day cycles
  Other Names: CGT9486; PLX9486
  Arms: (Part 1a) Bezuclastinib Dose 1 + BSC; (Part 1a) Bezuclastinib Dose 2 + BSC; (Part 3) Bezuclastinib + BSC
Drug: Bezuclastinib Tablets (Formulation B) — Bezuclastinib will be administered orally, once daily continuously for 28-day cycles
  Other Names: CGT9486; PLX9486
  Arms: (Part 1b) Bezuclastinib Dose 1 + BSC; (Part 1b) Bezuclastinib Dose 2 + BSC; (Part 2) Bezuclastinib Selected Dose + BSC; (Part 3) Bezuclastinib + BSC; (Prior Therapy Sub-study) Bezuclastinib
Drug: Placebo Tablets — Placebo will be administered orally, once daily continuously for 28-day cycles
  Arms: (Part 1a) Placebo + BSC; (Part 1b) Placebo + BSC; (Part 2) Placebo + BSC

SUMMARY:
This is a multi-part, randomized, double-blind, placebo-controlled Phase 2 clinical study comparing the safety and efficacy of bezuclastinib (CGT9486) plus best supportive care (BSC) with placebo plus BSC in patients with nonadvanced systemic mastocytosis (NonAdvSM), including indolent systemic mastocytosis and smoldering systemic mastocytosis, whose symptoms are not adequately controlled by BSC. This study will be conducted in three parts. Patients in Parts 1a, 1b and 2 will receive bezuclastinib or placebo, and may roll over onto Part 3 to receive treatment with bezuclastinib. Additionally, a substudy of subjects will investigate the efficacy, safety, and tolerability of bezuclastinib in patients who are experiencing inadequate symptom control with avapritinib.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosed with 1 of the following diagnoses according to the 2016 World Health Organization (WHO) classification for systemic mastocytosis (SM):

   * Indolent systemic mastocytosis (ISM),
   * Bone marrow mastocytosis (BMM)
   * Smoldering systemic mastocytosis (SSM)
2. Moderate-to-severe symptoms based on a minimum total symptom scoew (TSS) of the Mastocytosis Activity Score (MAS) and after establishing a stable regimen of at least 2 antimediator therapies over a 14-day eligibility period
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2
4. For patients receiving corticosteroids, the dose must be ≤10 mg/day of prednisone or equivalent

Key Exclusion Criteria:

1. Persistent toxicity from previous therapy for NonAdvSM that has not resolved to ≤ Grade 1
2. Diagnosed with any of the following WHO SM classifications: bone marrow mastocytosis, advanced systemic mastocytosis including SM with associated hematologic neoplasm, aggressive SM, mast cell leukemia; or mast cell sarcoma
3. Diagnosed with mastocytosis of the skin without systemic involvement
4. Received prior treatment with any targeted KIT inhibitor with the exception of approved agents for the treatment of SM
5. Received prior cytoreductive therapy or investigational agent for <14 days or 5 half- lives of the drug and for cladribine, interferon alpha, pegylated interferon, or antibody therapy <28 days or 5 half-lives of the drug (whichever is longer), before starting screening assessments
6. Received radiotherapy or psoralen and ultraviolet A therapy <14 days before starting screening assessments
7. Received any hematopoietic growth factor support <14 days or 5 half lives of the drug before starting screening assessments
8. History of clinically significant bleeding event within 30 days before the first dose of study drug or need for therapeutic anticoagulation on study
9. Need for treatment of corticosteroids at >10 mg/day of prednisone or equivalent
10. Received strong CYP3A4 inhibitors or inducers within 14 days or 5 drug half-lives before the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Part 1: Determine recommended dose of bezuclastinib (CGT9486) in subjects with NonAdvSM | 3 months
  Selection of the recommended dose to be used in subsequent parts of the study.
Part 2: Efficacy of bezuclastinib at the selected dose versus placebo | 24 Weeks
  Mean absolute change on the Mastocytosis Symptom Severity Daily Diary (MS2D2)
Part 3: Safety and tolerability of bezuclastinib as assessed by number of adverse events | Up to 5 years
  CTCAE v5

SECONDARY OUTCOMES:
Part 2: Proportion of subjects who had at least 50% reduction in serum tryptase | 24 weeks
Part 2: Proportion of subjects who had at least a 50% reduction in peripheral blood D816V allele fraction | 24 weeks
Part 2: Determine responder rates of subjects treated with bezuclastinib at the selected dose versus placebo | 24 weeks
  Proportion of subjects with at least a 30% reduction of the total symptom score (TSS) on the MS2D2.
  Proportion of subjects with at least a 50% reduction of the total symptom score (TSS) on the MS2D2.
Part 2: Proportion of subjects who had at least 50% reduction in mast cell burden | 24 weeks
Parts 1 & 2: Safety and tolerability of bezuclastinib as assessed by number of adverse events | Up to 24 weeks
  CTCAE v5
Parts 1, 2, & 3: Change and percent change in patient reported outcome (PRO) measures | Up to 5 years
Parts 1 & 3: Change and percent change in serum tryptase | Up to 12 months
Parts 1 & 3: Change and percent change in bone marrow mast cells | Up to 18 months
Part 1: Assess the pharmacokinetics (PK) of bezuclastinib in subjects with NonAdvSM | 3 months
  Plasma concentrations of CGT9846
Part 2: Determine mean change from baseline in predetermined PRO sub-domain and individual item scores | 24 weeks
Parts 2 & 3: Determine change of the lead (most severe) symptom and lead (most severe) subdomain of the MS2D2 in subjects treated with bezuclastinib versus placebo | Up to 5 years
  Change and percent change from baseline in the symptom score of the subject's most severe symptom.
  Change and percent change from baseline in the MS2D2 subdomain score of the subject's most severe subdomain.
Part 3: Change and percent change in the levels of KIT D816V mutation allele burden | Up to 12 months
Part 3: To determine the efficacy of bezuclastinib at the selected dose | Up to 2 years
  Proportion of subjects with at least a 50% reduction in MS2D2 TSS from baseline at 1 year and 2 years from start of bezuclastinib
  Change and percent change from baseline in the MS2D2 TSS, subdomain, and individual item scores
Part 3: Usage of concomitant medications as rescue therapy for NonAdvSM and changes from baseline in rescue therapy and best supportive care medications regimen | Up to 5 years

OTHER OUTCOMES:
Substudy: Efficacy of bezuclastinib at selected dose in subjects whose symptoms are not adequately controlled by avapritinib | Up to 2 years
  Mean absolute change on the Mastocytosis Symptom Severity Daily Diary (MS2D2)

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Easton, MD, PhD, Study Director — Cogent Biosciences
Locations (69):
- United States (29):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - One of a Kind Clinical Research Center, Scottsdale, Arizona
  - Modena Allergy and Asthma Clinical, La Jolla, California
  - University of California, Los Angeles (UCLA) - Medical Center, Los Angeles, California
  - Innovative Research of West Florida, Clearwater, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Allervie Clinical Research, Glenn Dale, Maryland
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Chesapeake Research Center, White Marsh, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic- Rochester, Rochester, Minnesota
  - Washington University at St. Louis, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University, Raleigh, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - AIR Care, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Metrodora Institute of Technology, West Valley City, Utah
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
- Austria (2):
  - Kepler Universitaetsklinikum GmbH, Linz
  - Medizinische Universitaet Wien, Vienna
- Belgium (2):
  - Antwerp University Hospital (UZA), Edegem
  - CHU Tivoli, La Louvière
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - St. Michael's Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- Fakultni nemocnice Kralovske Vinohrady, Prague, Czechia
- France (3):
  - AP-HM - Hopital de la Timone, Marseille
  - AP-HP- Hopital Pitie-Salpetriere, Paris
  - CHU de Toulouse - Hopital Larrey, Toulouse
- Germany (5):
  - Universitaetsklinikum Aachen, AoeR, Aachen
  - Charité Universitätsmedizin Berlin, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - University Medical Centre Mannheim, Mannheim
- Attikon University General Hospital Athens, Athens, Greece
- Ireland (2):
  - Cork University Hospital, Cork
  - St. James's Hospital, Dublin
- Italy (7):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - AOU Policlinico Rodolico San Marco, Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - AUSL della Romagna-Ospedale S.Maria delle Croci, Ravenna
  - Policlinico Universitario Agostino Gemelli, Rome
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale Borgo Trento, Verona
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Rotterdam, Rotterdam
- Oslo University Hospital, Oslo, Norway
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Klinika Hematologii i Transplantologii, Gdansk
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 - Klinika Hematoonkologii i Transplantacji Szpiku, Lublin
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Instituto de Estudios de Mastocitosis de Castilla La Mancha-Hospital Virgen del Valle, Toledo
- University Hospital Basel, Basel, Switzerland
- Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No